CLINICAL TRIAL: NCT06361147
Title: The Effect of Psychoeducation on Adult Siblings of People With Autism Spectrum Disorder.
Brief Title: Psychoeducation of Adult Siblings of ASD People (Autism Spectrum Disorder).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Mediterranean University (Other)
Responsible Party: Principal Investigator, Charalampos Depastas, PhD candidate in Social Work, Hellenic Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3764/2-10-2019
Record Dates: First submitted 2024-03-28; First posted 2024-04-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Sibling Relations
Keywords: psychoeducation; siblings; siblings relationship; ASD; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Interventional groups and Control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Psychoeducational program (group A - Ex. gr) (Experimental): This group of volunteers is going to participate in the online psychoeducational training program for ASD. Number of participants:11.
  To evaluate the effectiveness of the program, participants will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up).
  Interventions: Other: Psychoeducational program for ASD
- Psychoeducational program (group A - Co. gr) (No Intervention): Concurrently with the experimental group A, the no-interventional group will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up). Number of participants:11.
- Psychoeducational program (group Β - Ex. gr) (Experimental): This group of volunteers is going to participate in the online psychoeducational training program for ASD. Number of participants:11.
  To evaluate the effectiveness of the program, participants will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up).
  Interventions: Other: Psychoeducational program for ASD
- Psychoeducational program (group B - Co. gr) (No Intervention): Concurrently with the experimental group B, the no-interventional group will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up). Number of participants:11.
- Psychoeducational program (group C - Ex. gr) (Experimental): This group of volunteers is going to participate in the online psychoeducational training program for ASD. Number of participants:11.
  To evaluate the effectiveness of the program, participants will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up).
  Interventions: Other: Psychoeducational program for ASD
- Psychoeducational program (group C - Co. gr) (No Intervention): Concurrently with the experimental group C, the no-interventional group will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up). Number of participants:11.
- Psychoeducational program (group D - Ex. gr) (Experimental): This group of volunteers is going to participate in the online psychoeducational training program for ASD. Number of participants:11.
  To evaluate the effectiveness of the program, participants will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up).
  Interventions: Other: Psychoeducational program for ASD
- Psychoeducational program (group D - Co. gr) (No Intervention): Concurrently with the experimental group D, the no-interventional group will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up). Number of participants:11.

INTERVENTIONS:
Other: Psychoeducational program for ASD — 6 psychoeducation trainings for Autism Spectrum Disorder
  Arms: Psychoeducational program (group A - Ex. gr); Psychoeducational program (group C - Ex. gr); Psychoeducational program (group D - Ex. gr); Psychoeducational program (group Β - Ex. gr)

SUMMARY:
The aim of this study is to evaluate the effectiveness of a psychoeducational program in enhancing autism-related knowledge, sibling relationships, well-being, and resilience among adults with a sibling on the spectrum, while also highlighting the need for tailored supportive interventions for this population.

The psychoeducational program will be implemented in adult siblings of people with ASD and its effectiveness will be assessed.

Participation in this program is expected to contribute in the improvement of the quality of life of the participants, their siblings with ASD and those related to them. No risk is identified.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental lifelong disorder of which prevalence has been significantly increased through the decades. Notwithstanding the abundant research finding on the ASD people and their parents regarding their mental health, quality of life etc., limited evidence exists regarding the siblings of people with ASD. The aim of this study is to apply a psychoeducational program for ASD in adult siblings of people with ASD as a means of providing disorder - related knowledge and improving their quality of life. The psychoeducational program will provide basic knowledge about ASD, training on behavioral management, acceptance and ongoing support to serve the needs of people with ASD and their caregivers.

This study will be a randomized controlled trial (RCT) with voluntary participation. The psychoeducational program will be implemented in adult siblings of people with ASD, free of charge, it will be conducted online by certified trainers, due to the coronavirus pandemic and its effectiveness will be assessed. The sample will be recruited from the general population of Greece. Four groups, each divided into experimental groups and control groups, will be randomized.

To evaluate the effectiveness of the program, participants will be asked to complete the online questionnaires three times (pre-intervention, post-intervention and three-month follow-up).

Participation in this program is expected to contribute in the improvement of the quality of life of the participants, their siblings with ASD and those related to them. No risk is identified.

This study is part of a doctoral thesis in progress at the Hellenic Mediterranean University (HELMEPA), Department of Social Work.

The study is expected to start in April 2024 and to be completed about six months later.

ELIGIBILITY:
Inclusion criteria were: (i) age 18 or older, (ii) having one sibling diagnosed with ASD, (iii) being neurotypical, and (iv) no prior participation in a psychoeducational program for autism.

Exclusion criteria were: (i) having more than one sibling diagnosed with ASD, and (ii) residing outside Greece.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Psychoeducation effectiveness on the knowledge of ASD | 6 months
  The evaluation of psychoeducational program effect on knowledge of ASD is going to be evaluated throw the "Participatory Autism Knowledge Scale" questionnaire (29-item scale) will be used. The original validation studies demonstrated satisfactory psychometric properties, showing good internal consistency. The standardization and adaptation of the questionnaire into Greek has not yet been published in a peer-reviewed journal.
Psychoeducation effectiveness on siblings relationship | 6 months
  A newly developed research measure, designed specifically for this study to assess negative emotions and attitudes of adult siblings toward their autistic sibling. The questionnaire's name is "Adult Sibling Relationships and Autism Spectrum Questionnaire (ASRQ-AS) " - 31-item scale. The standardization and adaptation of the questionnaire into Greek has not yet been published in a peer-reviewed journal.
Psychoeducation effectiveness on resilience of siblings of ASD | 6 months
  The Brief Resilience Scale (BRS) was developed to assess an individual's ability to recover from stress and adversity. It can also be used to examine factors and outcomes associated with resilience in both mental and physical health, identifying individuals who may benefit from supportive or therapeutic interventions. The internal consistency (Cronbach's α) of the BRS demonstrates good reliability as well as in Greek version.
Psychoeducation effectiveness on the well-being of siblings of ASD | 6 months
  The evaluation of psychoeducational program effect on the well-being is going to be evaluated throw the questionnaire "PERMA-Profiler" (23-item scale). The scale has demonstrated adequate reliability and validity in assessing well-being - Cronbach's α values.

CONTACTS AND LOCATIONS:
Overall Officials: CHARALAMPOS DEPASTAS, PhD stud., Principal Investigator — Hellenic Mediterranean University
Locations (1):
- Hellenic Mediterranean University, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No
We will keep the anonymity of participants and there is no plan to share their data to other researchers.